CLINICAL TRIAL: NCT01610843
Title: Worldwide Sarcoidosis Research Study
Acronym: WISE
Status: Completed | Type: Observational
Sponsor: Alicia Gerke (Other)
Collaborators: National Center for Research Resources (NCRR) (NIH)
Responsible Party: Sponsor-Investigator, Alicia Gerke, Associate Professor; Division of Pulmonary, Critial Care and Occupational Medicine, University of Iowa
Organization: University of Iowa (Other)
Other Study IDs: 200907757; 5UL1RR024979 (NIH)
Record Dates: First submitted 2012-05-31; First posted 2012-06-04 (Estimated); Last update posted 2025-12-22 (Actual); Status verified 2025-12

CONDITIONS: Sarcoidosis
Keywords: Sarcoidosis; WISE; Sarcoid Study; Worldwide Sarcoidosis Research Study
MeSH Terms: conditions — Sarcoidosis | interventions — Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Saliva samples will be collected and processed at the University of Iowa.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Survey — Longitudinal surveys

SUMMARY:
The aim of this study is to collect information about the clinical course and characteristics of sarcoidosis patients around the world through web-based surveys. Recruitment is directed at and driven by patients in the sarcoidosis community. This will allow the the investigators to study sarcoidosis patients across all demographic, geographic, and socioeconomic boundaries, not just patients seen at large research centers. The investigators believe this study can give investigators a broader and less biased view of sarcoidosis. The investigators would also like to collect genetic samples on this population to assess genetic variance in different phenotypes.

The information for the study would be provided through a web based survey system that can be accessed by patients or physicians of patients from any computer with Internet access. This system would collect clinical information in sufficient detail so that the phenotype of individual patients can be evaluated. Upon agreeing to participate in further research studies through the website, subjects will also have the opportunity to provide a DNA sample.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of Sarcoidosis
* Access to a computer with Internet

Exclusion Criteria:

* None

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Individuals diagnosed with sarcoidosis who have a computer with Internet access.
Sampling Method: Non-Probability Sample
Enrollment: 2200 (Actual)
Dates: Start 2011-12 (Actual); Primary Completion 2025-07 (Actual); Study Completion 2025-10 (Actual)

PRIMARY OUTCOMES:
Define and characterize sarcoidosis phenotypes and methods of care | Anticipated by 2017
  To give a broader and less biased view of sarcoidosis

CONTACTS AND LOCATIONS:
Overall Officials: Alicia K Gerke, MD, Principal Investigator — University of Iowa
Locations (1):
- University of Iowa, Iowa City, Iowa, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Statement on sarcoidosis. Joint Statement of the American Thoracic Society (ATS), the European Respiratory Society (ERS) and the World Association of Sarcoidosis and Other Granulomatous Disorders (WASOG) adopted by the ATS Board of Directors and by the ERS Executive Committee, February 1999. Am J Respir Crit Care Med. 1999 Aug;160(2):736-55. doi: 10.1164/ajrccm.160.2.ats4-99. No abstract available. PMID 10430755
- [Background] Baughman RP, Teirstein AS, Judson MA, Rossman MD, Yeager H Jr, Bresnitz EA, DePalo L, Hunninghake G, Iannuzzi MC, Johns CJ, McLennan G, Moller DR, Newman LS, Rabin DL, Rose C, Rybicki B, Weinberger SE, Terrin ML, Knatterud GL, Cherniak R; Case Control Etiologic Study of Sarcoidosis (ACCESS) research group. Clinical characteristics of patients in a case control study of sarcoidosis. Am J Respir Crit Care Med. 2001 Nov 15;164(10 Pt 1):1885-9. doi: 10.1164/ajrccm.164.10.2104046. PMID 11734441
- [Background] Judson MA, Thompson BW, Rabin DL, Steimel J, Knattereud GL, Lackland DT, Rose C, Rand CS, Baughman RP, Teirstein AS; ACCESS Research Group. The diagnostic pathway to sarcoidosis. Chest. 2003 Feb;123(2):406-12. doi: 10.1378/chest.123.2.406. PMID 12576358
- [Background] Yeager H, Rossman MD, Baughman RP, Teirstein AS, Judson MA, Rabin DL, Iannuzzi MC, Rose C, Bresnitz EA, DePalo L, Hunninghakes G, Johns CJ, McLennan G, Moller DR, Newman LS, Rybicki B, Weinberger SE, Wilkins PC, Cherniack R; ACCESS Research Group. Pulmonary and psychosocial findings at enrollment in the ACCESS study. Sarcoidosis Vasc Diffuse Lung Dis. 2005 Jun;22(2):147-53. PMID 16053031
- [Background] Rybicki BA, Major M, Popovich J Jr, Maliarik MJ, Iannuzzi MC. Racial differences in sarcoidosis incidence: a 5-year study in a health maintenance organization. Am J Epidemiol. 1997 Feb 1;145(3):234-41. doi: 10.1093/oxfordjournals.aje.a009096. PMID 9012596
- [Background] Judson MA, Baughman RP, Thompson BW, Teirstein AS, Terrin ML, Rossman MD, Yeager H Jr, McLennan G, Bresnitz EA, DePalo L, Hunninghake G, Iannuzzi MC, Johns CJ, Moller DR, Newman LS, Rabin DL, Rose C, Rybicki BA, Weinberger SE, Knatterud GL, Cherniak R; ACCESS Research Group. Two year prognosis of sarcoidosis: the ACCESS experience. Sarcoidosis Vasc Diffuse Lung Dis. 2003 Oct;20(3):204-11. PMID 14620163
- [Background] Aranda A, Paramo JA, Rocha E. Fibrinolytic activity in plasma after gynecological and urological surgery. Haemostasis. 1988;18(2):129-34. doi: 10.1159/000215794. PMID 3137141
- [Background] Rabin DL, Thompson B, Brown KM, Judson MA, Huang X, Lackland DT, Knatterud GL, Yeager H Jr, Rose C, Steimel J. Sarcoidosis: social predictors of severity at presentation. Eur Respir J. 2004 Oct;24(4):601-8. doi: 10.1183/09031936.04.00070503. PMID 15459139
- [Background] Clark RE, McKnight RC, Kissane JM, Weldon CS. Experimentally reversed pulmonary blood flow. Implications for the surgical management of complex forms of congenital heart disease. Ann Thorac Surg. 1975 Oct;20(4):433-45. doi: 10.1016/s0003-4975(10)64241-5. PMID 1180597
- See also: Worldwide Sarcoidosis Research Study — http://www.sarcoidstudy.org